CLINICAL TRIAL: NCT02074748
Title: First Ray Kinematics Following Lapidus Bunion Surgery: A Fluoroscopic Gait Study
Brief Title: Measurement of Arch Motion After Bunion Surgery
Status: Terminated | Type: Observational
Why Stopped: Surgeons chose not to provide patients for testing
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Other Study IDs: 1401M47629
Record Dates: First submitted 2014-02-18; First posted 2014-02-28 (Estimated); Last update posted 2019-11-01 (Actual); Status verified 2019-10

CONDITIONS: Hallux Valgus; Instability of the Foot Arch
Keywords: Bunion; Foot Arch; Instability
MeSH Terms: conditions — Hallux Valgus; Bunion

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Bunion: Patients being treated for foot bunion with surgery.
- Controls (normal foot): Participants in this group will not undergo surgery.

SUMMARY:
This study is an observational "change from baseline" outcome measures design. Data is collected for the sake of evaluating treatment (fusion surgery) performed as standard medical care, but the investigator does not assign specific interventions to any participants in this study.

DETAILED DESCRIPTION:
Device/fluoroscopy measurements of arch motion and questionnaire data will be acquired on 10 women undergoing surgery for bunion, and 10 controls. Surgery will implant hardware to fuse (stabilize) the arch. Methods will evaluate the patient's problems associated with bunion and satisfaction with surgery, and assess the effectiveness of surgery in reducing motion of the arch. The hypotheses are that patients treated with surgery will demonstrate improvement in function, and that surgery will reduce motion of the arch postoperatively (posttest measures acquired 6 months after surgery), and in comparison to measures taken on a control group.

The data collected will come from a comprehensive examination. Methods will include the measurement of arch motion made by an examiner using a device and a fluoroscopic gait examination procedure, and completion of two medical questionnaires. The fluoroscopic acquisition of the digital images will be analyzed across the specified time dimensions of the gait cycle.

Device and fluoroscopy of measures of arch motion will be made at 2 time points on patients enrolled in this study: presurgery (baseline) and 6 months postsurgery. The questionnaire measurements of self-reported pain and function will be made at 4 time points: presurgery (baseline) and again at 3 months, 6 months, and 12 months postsurgery. Outcome measurements will be collected on control subjects at one time point only, on the day of their enrollment into the study.

Prospective studies have not characterized outcomes in patients receiving this type surgical fusion as part of the corrective treatment for bunion. Results have potential to improve surgical treatment outcomes and, improve upon the current methods of fluoroscopic motion analysis.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older.
* Women.
* Able to comprehend the risks associated with the study.
* Able to complete the paperwork required for enrollment.
* Able to walk without assistance of another individual.

Exclusion Criteria:

* Pregnancy
* History of great toe, forefoot or arch surgery, or severe traumatic injury.
* Reduced ankle or great toe motion that impairs the ability to walk.
* Observed evidence of foot deformity other than bunion.
* Insensate to skin sensation testing which could indicate neuropathy.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients having bunion will be recruited from the surgical practice of the Co-I. The surgeon will screen the patients, and invite those to participate identified as having an unstable arch as a complication of bunion deformity.
  Controls will be recruited from the community, group matched for age. Controls must have normal foot posture and display no evidence of an unstable arch.
Sampling Method: Non-Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2014-02; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Fluoroscopy Examination of the Foot. | Change in Outcome Measurement [presurgery (baseline) and again 6 months postsurgery]
  Fluoroscopic examination will image the foot during the roll-over phase of the gait. The participant will step in slow motion in front of the fluoroscopic x-ray beam to record the change in the position of the arch at specified gait-event time dimensions. Image acquisition will be at 25 frames per second lasting no longer than 2 seconds. All participants will wear leaded clothing in accordance with a protocol approved by the Univ of Minnesota Department of Health and Safety, Radiation Protection Division.
  Fluoroscopy "change in outcome measures" of arch motion will be made at 2 time points on all patients who participate: presurgery (baseline) and again 6 months postsurgery.
  Fluoroscopy measures will be acquired on control subjects at one time point only, on the day of their enrollment into the study.

SECONDARY OUTCOMES:
Device Measurement of Arch Motion. | Change in Outcome Measurement. [presurgery (baseline) and again 6 months postsurgery]
  Device measurement of arch motion will be acquired using the device built for this one purpose. Device measurements will be made on the both feet.
  Device "change in outcome measurement" of arch motion will be made a 2 time points on all patients: presurgery (baseline) and again 6 months postsurgery.
  Device measures of arch motion will be acquired on control subjects at one time point only, on the day their enrollment into the study.

OTHER OUTCOMES:
Medical Questionnaires. | Change in Outcome Measurements. [presurgery (baseline) and again at 3 months, 6 months, and 12 months postsurgery]
  The Foot Function Index medical questionnaire has separate subscales that assess health in the multiple dimensions of pain, activity limitation, disability and stiffness. Level of pain will also be recorded on the standard 1-10 medical pain scale.
  The "change in outcome measures" of the self-reported pain and function will be made at 4 time points on all patients who participate: presurgery (baseline) and again at 3 months, 6 months, and 12 months postsurgery.
  Questionnaire measures will be acquired on control subjects at one time point only, on the day of their enrollment into the study.

CONTACTS AND LOCATIONS:
Overall Officials: Ward M Glasoe, PhD, PT, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States